CLINICAL TRIAL: NCT00548821
Title: A Phase III Randomized Trial Between 5 Day 3 Weekly and Weekly Cisplatin Based Chemotherapy for Patients With Locally Advanced Cervical Cancer
Brief Title: Randomized Trial Between Weekly and 5 Day 3 Weekly Cisplatin for Cervical Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Dr Johann Tang, National University Hospital, Singapore
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cervix Cancer Research
Record Dates: First submitted 2007-10-23; First posted 2007-10-24 (Estimated); Last update posted 2008-05-15 (Estimated); Status verified 2008-05

CONDITIONS: Locally Advanced Cervical Cancer
MeSH Terms: interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Experimental): ARM 2: Weekly cisplatin 40mg/m2, concurrent with radiotherapy.
  Interventions: Drug: Cisplatin
- 1 (Experimental): ARM 1: 5-day 3 weekly cisplatin 20mg/m2 for 5 days, concurrent with radiotherapy
  Interventions: Drug: Cisplatin

INTERVENTIONS:
Drug: Cisplatin

SUMMARY:
The primary aim of this research protocol is to compare if there is a difference in progression free survival between weekly versus 5-day 3 weekly cisplatin based chemotherapy regimen in women with locally advanced cervical cancer. The secondary aims are to compare quality of life assessment of patients and their carers as well as toxicity profiles both acute and late.

ELIGIBILITY:
Inclusion Criteria:

* stage IB2-IVA , histological proven cervical carcinoma
* no previous diagnosis of carcinoma
* no prior history of chemotherapy or radiotherapy
* ECOG less than or equal to 2
* Above 21 years old
* medically fit for radical concurrent Cisplatin based chemotherapy and radiotherapy
* Hemoglobin >10g/dL
* Adequate hematological, renal and hepatic function according to all of the following laboratory values:

  * Absolute neutrophil count ≥ 1.5 ×109/l
  * Platelets ≥ 100 ×109/l
  * Serum creatinine ≤ 1.5 times upper limit of laboratory normal
  * Total serum bilirubin ≤ 1.5 times upper limit of laboratory normal
  * ASAT(AST) or ALAT(ALT) ≤ 2.5 times upper limit of laboratory normal
  * Alkaline phosphatase of ≤ 2.5 times upper limit of laboratory normal

Exclusion Criteria:

* Age below 21
* Presence of known HIV infection, chronic hepatitis B or hepatitis C infection
* Psychological, familial, sociological, or geographical condition that would preclude study participation
* Prior (within the last 3 years) or simultaneous malignancies (other then cutaneous basal cell carcinoma or non-invasive tumors)
* Patients with the following histologies are excluded: small cell, carcinoid, glassy cell, clear cell and adenoid cystic.
* Life expectancy < 6 months
* Patients with insulin dependent diabetes
* Prior tumor-directed surgery
* Previous systemic chemotherapy or pelvic radiation therapy
* As radiation and cytotoxic agents are contraindicated in pregnancy, pregnant women are ineligible and those of childbearing potential should use contraception

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
The primary aim of this research protocol is to compare if there is a difference in progression free survival between weekly versus 5-day 3 weekly cisplatin based chemotherapy regimen in women with locally advanced cervical cancer.

SECONDARY OUTCOMES:
The secondary aims are to compare quality of life assessment of patients and their carers as well as toxicity profiles both acute and late.

CONTACTS AND LOCATIONS:
Overall Officials: Johann Tang, Principal Investigator — NUH
Locations (1):
- National University Hospital, Singapore, Singapore